CLINICAL TRIAL: NCT04808739
Title: Retrospective Observational Study to Analyze the Effectiveness of Adalimumab
Brief Title: Adalimumab Biosimilar in Clinical Practice
Status: Completed | Type: Observational
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Other Study IDs: IIBSP-ADA-2020-32
Record Dates: First submitted 2021-03-17; First posted 2021-03-22 (Actual); Last update posted 2021-03-22 (Actual); Status verified 2021-03

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — Adalimumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: Adalimumab — Analysis of survival of adalimumab biosimilar in clinical practice

SUMMARY:
This is an observational, retrospective, multicenter, and descriptive study of patients treated with adalimumab biosimilar for psoriasis, according to clinical practice.

Existing data will be collected from the Dermatology Services database of the hospitals participating in the study, from the medical histories of all treated patients who meet the inclusion criteria and sign informed consent.

The aim of the study is to determine the effectiveness of the different adalimumab biosimilars in clinical practice.

DETAILED DESCRIPTION:
Adalimumab is indicated for the treatment of moderate to severe chronic plaque psoriasis in adult patients who are candidates for systemic treatment. There are currently several biosimilar drugs (Amgevita, Imraldi, Hyrimoz, Idacio, Hulio,…) in addition to the reference product (Humira).

The reduction in the cost of production of biosimilar drugs with respect to reference products has led to their replacement by biosimilar drugs in patients initiating biological therapy, but some centers are also switching to adalimumab biosimilar in patients who are controlled with original adalimumab (Humira).

There are no actual clinical efficacy / safety data in our setting on the use of adalimumab biosimilars.

There is also no evidence of maintenance response in patients who are switched from adalimumab (Humira) to biosimilar adalimumab in clinical practice.

This retrospective study will collect demographic and disease data of the psoriasis patient treated with the different biosimilars of adalimumab, as well as their comorbidities, response to treatment, and safety. In this way, data will be available in usual clinical practice to improve the management of the patient with psoriasis treated with biosimilar drugs.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes who have received treatment with adalimumab and who have signed an informed consent.

Exclusion Criteria:

* Refusal to participate.
* Any other cause of exclusion based on clinical criteria and the technical data sheet of the drug.

Ages: 2 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with moderate-severe psoriasis vulgaris who are candidates for systemic treatment undergoing adalimumab treatment.
Sampling Method: Non-Probability Sample
Enrollment: 604 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
Median time of survival (months) of adalimumab biosimilar in clinical practice | 1 year
  Median time of survival (months) of patients under treatment with adalimumab biosimilar in clinical practice

CONTACTS AND LOCATIONS:
Overall Officials: Lluís Puig, MD, PhD, Principal Investigator — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau
Locations (1):
- Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No
IPD will be collected and data analysed in Institut de Recerca Hospital de la Santa Creu i Sant Pau

REFERENCES:
- [Background] Khandpur S, Sondhi P, Taneja N, Sharma P, Das D, Sharma A, Sreenivas V. Evaluation of adalimumab biosimilar in treatment of psoriatic arthritis with concomitant moderate to severe chronic plaque psoriasis: An open-labeled, prospective, pilot case series. J Am Acad Dermatol. 2020 Jul;83(1):248-251. doi: 10.1016/j.jaad.2019.12.071. Epub 2020 Feb 19. No abstract available. PMID 32087993
- [Background] Reynolds KA, Pithadia DJ, Lee EB, Liao W, Wu JJ. Safety and Effectiveness of Anti-Tumor Necrosis Factor-Alpha Biosimilar Agents in the Treatment of Psoriasis. Am J Clin Dermatol. 2020 Aug;21(4):483-491. doi: 10.1007/s40257-020-00507-1. PMID 32048187
- [Background] Hercogova J, Papp KA, Chyrok V, Ullmann M, Vlachos P, Edwards CJ. AURIEL-PsO: a randomized, double-blind phase III equivalence trial to demonstrate the clinical similarity of the proposed biosimilar MSB11022 to reference adalimumab in patients with moderate-to-severe chronic plaque-type psoriasis. Br J Dermatol. 2020 Feb;182(2):316-326. doi: 10.1111/bjd.18220. Epub 2019 Sep 26. PMID 31206593